CLINICAL TRIAL: NCT06038487
Title: Immediate Versus Delayed Loading of Maxillary Overdenture Implants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: Institut Straumann AG (Industry)
Responsible Party: Principal Investigator, Gian Schincaglia, Professor, Chair and Graduate Program Director, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY20221174
Record Dates: First submitted 2023-09-08; First posted 2023-09-14 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Implant Complication
Keywords: Implant Overdenture; Immediate loading; Delayed loading; Maxillary Overdenture; Novaloc Retention System; Guided Implants; Immediate vs Delayed loading; Implant-supported overdenture

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Masking Description: Every patient will be given a participant identification number. An independent investigator, not involved with patient treatment, will generate the allocation list. Computer software will be used to randomize the participant identification numbers into one of the two groups. This information will be concealed in sealed opaque envelopes, which will be open after implants are placed. Neither the surgeon, nor the patient will be aware of the group assignment until after implant insertion.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test - IL ( Immediate Loading) (Experimental): The maxillary denture will be immediately connected to the implants on the day of the surgery
  Interventions: Procedure: Immediate loading of maxillary implant overdenture
- Control - DL ( Delayed Loading) (Active Comparator): At the time of surgery, the cover screw will be seated on the implants and the flap will be sutured for a submerged healing. After 3 months of healing the implants will be exposed and connected to the prosthesis following the same prosthetic protocol as the test group.
  Interventions: Procedure: Delayed loading of maxillary implant overdenture

INTERVENTIONS:
Procedure: Immediate loading of maxillary implant overdenture — The denture will be immediately connected to the implants. The abutment screw will be torqued at 15 Ncm. The Novaloc cap attachments will be picked up intra-orally using cold curing resin. To avoid contact of the resin with the surgical wound, a circular portion of a sterile rubber dam sheet will be adapted on the cap attachment once placed on the abutment during the pickup procedure. Occlusion is then checked and adjusted if necessary as well as the adaptation on the residual ridges and the patient dismissed. The patients in the test group will be instructed not to remove the prosthesis for one week.
  Arms: Test - IL ( Immediate Loading)
Procedure: Delayed loading of maxillary implant overdenture — A cover screw will be seated on the implants and the flap will be sutured for a submerged healing. After 3 months of healing the implants will be exposed and connected to the prosthesis following the same prosthetic protocol as described for the test group. The abutment screw will be torqued at 35 Ncm. As post-surgical instructions, the patients will be asked not to brush the operated areas and to rinse instead with 0,12% chlorhexidine solution twice a day for 1 minute for 14 days. Pain control is provided with 400 mg ibuprofen, as needed. Soft diet is recommended for 2 weeks. The patients in the control group will be asked not to wear the denture for 7 days.
  Arms: Control - DL ( Delayed Loading)

SUMMARY:
The purpose of the study is to evaluate the radiographic, clinical and patient-centered outcomes of implant-retained immediately-loaded maxillary complete dentures in comparison to delayed loading approach by primarily evaluating radiographic bone loss of dental implants placed in the maxilla over 36 months

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate radiographically at 6, 12, 24, and 36 months post-loading the performance of the BLX Roxolid™ implants placed using a flapless guided surgery and immediately loaded with a maxillary overdenture versus delayed loading 3 months after surgical placement. The outcome will be evaluated using peri-implant, radiographic bone level changes from baseline to 6, 12, 24, and 36 months post-implant placement. The secondary objectives include evaluation of the condition of the peri-implant mucosa (pocket depth and bleeding on probing); Implant survival at 6, 12, 24, and 36 months; The nature and the frequency of surgical and prosthetic complications; Patient-centred outcomes (OHIP 14). An initial evaluation will be conducted to determine whether a patient meets the study inclusion criteria. This evaluation will include medical history, clinical examination, and radiographic examination (OPT). A pre-operative prosthetic evaluation of the existing prostheses will be made to establish their quality and the need for a new set of complete dentures before the implant placement. The maxillary denture will be used as a radiographic guide for the pre-treatment CBCT assessment. The tridimensional image obtained with the CBCT will be used for the surgical planning of the implant positioning using a dedicated implant planning software (coDiagnostix, Dental Wings Gbmh, Chemniz Germany) and a stereo-lithographic surgical guide will obtained using a 3D printer (Formlab 3B, Formlabs Inc. Somerville MA.). The implants will be inserted under local anesthesia, following consumption of prophylactic antibiotic medications consisting of 2 grams of amoxicillin 1 hour before the surgical procedure. If the patient is allergic to penicillin or penicillin derivatives, azithromycin or other classes of antibiotics will be administered according to ADA guidelines. The implant placement will be performed using the stereo-lithographic surgical guide. A small crestal incision and a minimal flap elevation will be performed in the location of the implant sites. The osteotomy site will be prepared following the drilling sequence provided by the manufacturer's surgical manual. The implant will be placed, and the maximum value of insertion torque (peak of insertion torque, IT) will be measured during the seating of the most coronal implant threads using the surgical unit (W&H, Burmoos, Austria) and recorded as 20, 30, 40, 50 N/cm IT category. In case of IT lower than 20 N/cm the patient will be excluded from the study and the implant treatment will be completed following the standard delayed protocol. After implant placement, the patient will be randomly allocated to the test or control group. BLX Roxolid dental implants will be used, and length and size will be chosen based on the available bone volume. A minimum amount of bone at the 2nd premolar position to house a 3.5 x 10 mm BLX-Roxolid will be required. The patient will be randomly assigned to have their implants immediately loaded or conventionally loaded/delayed. The randomization will be computer-generated and the subject's assignment will be placed in a sealed envelope. On the day of surgery, after the implants are placed, the investigators will open the envelope to see which group the patient has been assigned to. If assigned to the test group, the denture will be immediately connected to the implants. The abutment screw will be torqued at 15 Ncm. The Novaloc cap attachments will be picked up intra-orally using cold-curing resin. To avoid contact of the resin with the surgical wound, a circular portion of a sterile rubber dam sheet will be adapted on the cap attachment once placed on the abutment during the pickup procedure. Occlusion is then checked and adjusted if necessary as well as the adaptation on the residual ridges and the patient is dismissed. If assigned to the control group, a cover screw will be seated on the implants and the flap will be sutured for submerged healing. After 3 months of healing the implants will be exposed and connected to the prosthesis following the same prosthetic protocol as described for the test group. The abutment screw will be torqued at 35 Ncm. As per post-surgical instructions, the patients will be asked not to brush the operated areas and to rinse instead with 0,12% chlorhexidine solution twice a day for 1 minute for 14 days. Pain control is provided with 400 mg ibuprofen, as needed. A soft diet is recommended for 2 weeks. The patients in the test group will be instructed not to remove the prosthesis for one week. The patients in the control group will be asked not to wear the denture for 7 days. Patients will be recalled at 1, 2, 4, 12 weeks, and 6, 12, 24, and 36 months after surgery. At the post-operative visit occlusion will be checked, as well as stability and retention of the prostheses and the need for any prosthetic maintenance. At 12 weeks the test group patient will have the abutment screw torqued at 35 Ncm. The control group patient will have the implant exposed and connected to Novaloc using a 35 Ncm torque. Periapical radiographs will be taken at abutment connection and 6, 12, 24, 36 months visit by paralleling technique using a Rinnâ (Dentsply Rinn, Elgin, Illinois, USA) film holder. The film holder will be indexed on the attachment so that the film position can be reproduced for the follow-up radiographs. All patient complaints or any complications resulting from a change in health status from baseline or any implant-related complications such as pain, paraesthesia, or peri-implant infection will be recorded as an adverse event in the CRF and will be monitored until the condition is resolved. OHIP-14 questionnaire will be administered at baseline, at 4 weeks post-surgery, and months 6, 12, 24, and 36 months.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females must be at least ≥ 21 years of age
2. Fully edentulous maxilla
3. The implant site has to be healed for at least 4 months after extraction
4. Wearing complete dentures deemed adequate
5. Orthopantomogram available (OPT)
6. Adequate amount of bone at least at the 2nd premolar position to house at minimum a 3.5 x 10 mm BLX-Roxolid implant
7. No bone grafting required
8. Implant IT ≥ 20 N/cm

Exclusion Criteria:

1. Conditions requiring chronic routine prophylactic use of antibiotics
2. Conditions requiring prolonged use of steroids
3. History of leukocyte dysfunction and deficiencies
4. Bleeding disorders
5. History of neoplastic disease requiring use of radiation or chemotherapy
6. Metabolic bone disorders
7. Uncontrolled endocrine disorder
8. Use of any investigational drug or device within the 30-day period prior to implant surgery
9. Vaping, Tobacco Chewing or Smoking more than 10 cigarettes a day
10. Alcoholism or drug abuse
11. Patient infected with HIV
12. Condition or circumstances, in the opinion of the investigator, which would prevent completion of study participation or interfere with analysis of study results, such as as history of non-compliance, unreliability.
13. Local inflammation including untreated periodontitis
14. Mucosal disease such as erosive lichen planus
15. History of local irradiation therapy
16. Osseous lesion
17. Severe bruxism and clenching habits
18. Active infection with suppuration or fistula track
19. Persistent intraoral infection
20. Lack of primary stability <20Ncm. In this instance, the patient must be withdrawn and treated according to the standard protocol.
21. Inadequate oral hygiene or unmotivated home care.
22. Bone grafting needed
23. Inadequate bone volume for implants insertion as measured on the pre-treatment cone beam computed tomography (CBCT).

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Radiographic bone level of changes of implants | 36 months
  The primary objective of this study is to evaluate radiographically at 6, 12, 24 and 36 months post-loading the performance of the BLX Roxolid™ implants placed using a flapless guided surgery and immediately loaded with a maxillary overdenture versus delayed loading 3 months after surgical placement. The outcome will be evaluated using peri-implant, radiographic bone level changes measure in milimeters from standardized radiographs from baseline to 6, 12, 24 and 36 months post implant placement.

SECONDARY OUTCOMES:
Pocket Depth of the peri-implant mucosa | 36 months
  Will be recorded as a whole number in milimeters at 6 sites per implant
Bleeding on probing of the peri-implant mucosa | 36 months
  Will be recorded as a absence or presence of bleeding on probing at 6 sites per implant
Implant survival | 36 months
  Implant survival at 6, 12, 24 and 36 months will be recorded as implant present or implant lost
Complications | 36 months
  The nature of surgical and prosthetic complications. For example, fracture of denture or loosening of implant abutment.
Patient-centered outcomes | 36 months
  Patient-centered outcomes according to Oral Health Impact Profile-14 (OHIP 14). The subjects will answer questions about their dentures and the potential problems they encounter and will have answer options of "very often," "fairly often," "occasionally," "hardly ever," "never," or "don't know." "Never" is considered the best outcome

CONTACTS AND LOCATIONS:
Overall Officials: Gian P Schincaglia, DDS, PhD, Principal Investigator — Case Western Reserve University
Locations (1):
- Case Western Reserve University Department of Periodontics, Cleveland, Ohio, United States

DOCUMENTS (1):
  • Informed Consent Form (2023-03-17): https://cdn.clinicaltrials.gov/large-docs/87/NCT06038487/ICF_000.pdf